CLINICAL TRIAL: NCT06305624
Title: Implementation of Mobile-based Programs for Alcohol Cessation in Treatment of Alcohol-associated Liver Disease (IMPACT-ALD): Aim 1
Brief Title: Implementation of Mobile-based Programs for Alcohol Cessation in Treatment of Alcohol-associated Liver Disease
Acronym: IMPACT-ALD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0130; 1R01AA030470-01A1 (NIH); A532000 (Other: UW Madison); Protocol Version 2/2/25 (Other: UW Madison)
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder; Alcohol-related Liver Disease
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, Type 1 hybrid implementation-effectiveness trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connections App (Experimental): The Connections app is based on principles of effective care for substance use disorders, such as sustained duration, peer support, improving coping skills in high-risk situations, assertive outreach, self- monitoring, prompts, and action planning. The theoretical foundation of CHESS Health is self-determination theory, which holds that an individual's adaptive functioning can be improved if the patient feels (1) competent, (2) related to others, and (3) internally motivated rather than coerced in one's actions.
  Interventions: Device: Connections App
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Device: Connections App — mobile application, a place where participants can find community and support to help them manage their ALD, learn liver health self-care, coping skills, and alcohol abstinence strategies.
  Arms: Connections App

SUMMARY:
This protocol describes a randomized controlled trial testing the effectiveness and implementability of the CHESS Health Connections smartphone application among patients with alcohol-associated liver disease (ALD) at two medical centers in Michigan and Wisconsin, in two types of clinics: general hepatology and multidisciplinary that offers care for advanced ALD alongside co-located, integrated mental health and substance abuse treatment. The long-term goal of this and future work is to prevent disease progression and promote healthy behaviors by improving the rate of abstinence among patients with ALD earlier in the course of their disease. 298 participants will be enrolled and can expect to be on study for up to 6 months.

DETAILED DESCRIPTION:
The goal of this project is to implement and evaluate an evidence-based mHealth system to help patients diagnosed with ALD with alcohol cessation. Connections is a mobile health app developed by CHESS Health to support patients with alcohol use disorders. Patients will be enrolled in both general hepatology and multidisciplinary ALD clinics (which include integrated alcohol use treatment professionals alongside hepatology providers) at two large tertiary care centers (University of Wisconsin (UW) and University of Michigan (UM)). The hypothesis is that the implementation of an adapted version of Connections for patients with ALD will improve rates of alcohol cessation and improve liver function.

* Aim 1 (described in this record) will assess the effectiveness of the Connections app plus usual care (n=149) compared to usual care (n=149) on days of alcohol abstinence over 6 months.
* Aim 2 will assess the implementation of the Connections app through qualitative interviews of key patient, provider, and clinic-level stakeholders using the Replicating Effective Programs framework. Aim 2 follows the study intervention phase and is not part of this record.

Secondary analyses will examine use of the Connections app on health outcomes (including depression, anxiety, insomnia, liver health, and quality of life) and health behaviors (including engagement with alcohol use disorder (AUD) and/or ALD treatments and ongoing alcohol use). Key moderators (including age, sex, race, ethnicity, marital status, rurality, and ALD severity) and mediators (including relatedness, competence, autonomous motivation) on outcomes will be explored. The impact of the Connections app on measures of chronic liver impairment documented in the health record will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALD (any stage)
* Alcoholic liver disease (ALD) encompasses a spectrum of hepatic injuries caused by long-term alcohol abuse. For this study, participants will have a diagnosis of ALD.
* Alcohol use within the last 6 months
* Receiving care at UW or Henry Ford Health + MSU

  * Either the general hepatology clinic or the multidisciplinary ALD clinic
* Able to read and write proficiently in English
* Willing and able to use a smartphone app

Exclusion Criteria:

* Actively listed for liver transplant or history of liver transplant before being enrolled in the study. Participants added to a liver transplant list after being enrolled in the study will be allowed to continue their participation
* In hospice care
* Has severe cognitive impairment (as described in electronic health record including dementia, delirium, and/or unable to maintain cognitive alertness during screening--as determined by study staff.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Days of Alcohol Abstinence in ALD Participants | data collected monthly, up to 6 months
  Alcohol consumption outcomes will be collected monthly and include whether or not alcohol was consumed on each of the past 30 days. Alcohol consumption outcomes will be compared between the usual care condition and the usual care plus the Connections app condition.
Number of Standard Drinks Consumed in ALD Participants | data collected monthly, up to 6 months
  Alcohol consumption outcomes will be collected monthly and include whether or not alcohol was consumed on each of the past 30 days, if yes, participant's will also be asked the number of standard drinks for each day alcohol was consumed. Alcohol consumption outcomes will be compared between the usual care condition and the usual care plus the Connections app condition.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-8) Score | baseline, 3 months, 6 months
  The PHQ-8 score is a measure of depressive symptoms that ranges from 0 to 24 where higher scores indicate increase depression.
Change in PROMIS Global Health Score | baseline, 3 months, 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Score is a measure of quality of life. It is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health Score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Change in Generalized Anxiety Disorder (GAD-7) Score | baseline, 3 months, 6 months
  GAD-7 is a measure of anxiety and has a range of scores from 0-21 where higher scores indicate increased anxiety.
Change in Insomnia Severity Index (ISI) Score | baseline, 3 months, 6 months
  ISI is a measure of insomnia and has a range of scores from 0-28 where higher scores indicate increased insomnia.
Change in Pain Interference (PEG) Score | baseline, 3 months, 6 months
  PEG is a pain measure scored from 0 (no pain or interference) to 10 (worst pain and complete interference).
Change in Drinking Motivations Questionnaire - Adult (DMQ-A) Score | baseline, 3 months, 6 months
  DMQ-A is a measure of drinking motivations, scored from 1-5 in each of 5 domains: social, coping, confidence, taste, enhancement. Higher scores indicate higher motivation to drink.
Change in CHESS Bonding Scale Score | baseline, 3 months, 6 months
  The CHESS Bonding Scale is an adapted measure developed to "capture the concept of universality, group cohesiveness, and informational and emotional support". Score from 0 to 20 where higher scores indicates increased bonding.
Change in Drug-Taking Confidence Questionnaire (DTCQ-8A) Score | baseline, 3 months, 6 months
  DTCQ-8A is a measure of self-efficacy scored from 0-100 where higher scores indicate greater self-efficacy.
Change in Treatment Self-Regulation Questionnaire (TSRQ) Score | baseline, 3 months, 6 months
  TSRQ is a measure of self-regulation scored from 1 to 7 in each of 4 domains: autonomous motivation, introjected regulation, external regulation, amotivation. Higher scores indicate more self-regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Quanbeck, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Henry Ford + Michigan State University Health Center, Lansing, Michigan
  - UW General Hepatology Clinic, Madison, Wisconsin
  - UW Multidisciplinary ALD Clinic, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Participant-level data that have been de-identified will be deposited and made available in a data repository maintained by NIAAA and referenced as NIAAA-DA. The National Institute on Alcohol Abuse and Alcoholism Data Archive (NIAAADA) is a data repository that houses and shares human subjects' data generated by NIAAA-funded research.
  Data released through NIAAA-DA are assigned a citation that includes a Global Unique Identifier (GUID). The GUID is a unique persistent identifier maintained by NIAAA-DA to ensure the data can be permanently identified. The citation and GUID are available on the study page and are provided with each download.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared with the general research community at the time of an associated outcomes publication, or the end of the award/support period, whichever comes first. Data will be retained in NIAAA-DA for the life of the repository.